CLINICAL TRIAL: NCT01371370
Title: Effects of Low-intensity Resistance Exercise Training and Diet on Central Hemodynamics and Arterial Stiffness in Obese Middle-aged Women With High Blood Pressure
Brief Title: Low-intensity Resistance Exercise and Diet on Arterial Function and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Nutrisystem, Inc. (Industry)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011.5485
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Pre-hypertension; Hypertension
Keywords: low intensity resistance exercise training; hypocaloric diet; prehypertension; hypertension; obesity; arterial function; arterial stiffness; pulse wave velocity; autonomic function; endothelial function; adipocytokines
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension | interventions — Resistance Training; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Resistance exercise training (Experimental): Lower-body exercises 3 times per wk for 12 wk
  Interventions: Other: Resistance exercise training
- Hypocaloric diet (Experimental): This arm involves 12 wk of the standard Nutrisystem foods plan complemented by fresh produce and dairy. Subjects consume breakfast, lunch, dinner, and one (women) or two (men) snacks per day.
  Interventions: Other: Hypocaloric diet
- Resistance exercise training & diet (Experimental): Lower-body exercise training and diet
  Interventions: Other: Resistance exercise training & diet
- Control (No Intervention): This arm involves not making any change to the subject's lifestyle at the moment of the start of the intervention and for 12 wk.

INTERVENTIONS:
Other: Resistance exercise training — The low intensity resistance exercise training intervention consists of lower-body resistance exercise (machines) 3 times per wk for 12 wk. Two sets the first 2 wk and 3 sets the rest of the intervention, at 40% of the estimated 1 repetition maximum, for 17 to 23 repetitions, with 1 minute of rest in between sets.
  Arms: Resistance exercise training
Other: Hypocaloric diet — The hypocaloric diet intervention consists of 12 wk of the standard Nutrisystem foods plan complemented by fresh produce and dairy. Subjects consume breakfast, lunch, dinner, and one (women) or two (men) snacks per day.
  Arms: Hypocaloric diet
Other: Resistance exercise training & diet — Combination of low intensity resistance exercise training and hypocaloric diet
  Arms: Resistance exercise training & diet

SUMMARY:
* Obesity is a major risk factor for premature arterial abnormalities including high blood pressure and increased stiffness. Previous studies have shown that weight loss via lifestyle modifications is associated with a decrease in large artery (aorta) stiffness. However, along with decreases in fat mass, hypocaloric diet reduces muscle mass. Low-intensity resistance exercise training (LIRET) results in similar increases in muscle mass and strength than those observed after high-intensity resistance exercise.
* The investigators hypothesis is that weight loss via diet combined with LIRET would additively reduce arterial stiffness and blood pressure (BP) in obese women. The investigators also hypothesize that the improved arterial function with weight loss would be associated with beneficial changes in the main mechanisms involved in BP regulation.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effects of 12 weeks of low-intensity resistance exercise training (LIRET) and diet on arterial function, autonomic function, and body composition in obese women with high blood pressure (BP). Specific aims of the study are to:

* To evaluate the extent to which diet and LIRET will improve body composition assessed by changes in fat mass and lean mass using dual-energy x-ray absorptiometry and waist circumference.
* To investigate that combined diet and LIRET are more efficacious than either treatment alone in ameliorating cardiovascular disease risk factors by assessing arterial stiffness (aortic, systemic, and leg), aortic BP and wave reflection, and autonomic function (heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and baroreflex sensitivity). Circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NO metabolites [NOx] and prostacyclin) and vasoconstrictors (endothelin-1 and prostaglandin F2α) will be assessed as secondary outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40 to 65 years of age
* Body mass index of 27-39.9
* Sedentary or low active (less than 2 hr per wk)

Exclusion Criteria:

* Younger than 40 or older than 65 years of age
* Body mass index lower than 27, or 40 or higher
* Physically active or competitively active
* Smoker
* Systolic blood pressure higher than 140 mmHg
* Use of hormone replacement therapy of less than 1 yr
* Use of calcium channel blocker or beta blockers
* Type 1 diabetes
* Uncontrolled type 2 diabetes

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 12 weeks
  Non-invasive measures of brachial and aortic blood pressure

SECONDARY OUTCOMES:
Autonomic Function | 12 weeks
  Heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and spontaneous baroreflex sensitivity will be assessed from electrocardiogram and beat-by-beat digital blood pressure
Endothelial Function | 12 weeks
  By measuring circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NO metabolites [NOx] and prostacyclin) and vasoconstrictors (endothelin-1 and prostaglandin F2α)
Body Composition | 12 weeks
  By measuring fat mass and lean soft tissue mass from dual-energy x-ray absorptiometry and waist circumference
Arterial Stiffness | 12 weeks
  Using pulse wave velocity of the aorta, systemic, and legs
Pressure Wave Reflection | 12 weeks
  Using the augmentation index from radial tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, M.D., Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Figueroa A, Vicil F, Sanchez-Gonzalez MA, Wong A, Ormsbee MJ, Hooshmand S, Daggy B. Effects of diet and/or low-intensity resistance exercise training on arterial stiffness, adiposity, and lean mass in obese postmenopausal women. Am J Hypertens. 2013 Mar;26(3):416-23. doi: 10.1093/ajh/hps050. Epub 2013 Jan 7. PMID 23382493